CLINICAL TRIAL: NCT00344214
Title: Reducing HIV/STD Risk, Methamphetamine Use, and Depression Among Heterosexuals
Brief Title: STD Risk Reduction for Heterosexual Methamphetamine Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Thomas L. Patterson, Professor in Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH061146 (NIH); R01MH061146 (NIH); DAHBR 9A-ASPQ
Record Dates: First submitted 2006-06-23; First posted 2006-06-26 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-09

CONDITIONS: Substance-Related Disorders; HIV Infections; Sexually Transmitted Diseases
Keywords: HIV; STDs; Methamphetamine
MeSH Terms: conditions — Substance-Related Disorders; HIV Infections; Sexually Transmitted Diseases | interventions — Standard of Care

ARMS (2):
- 1 (Experimental): Participants will receive the tri-focal cognitive behavioral therapy - social skills training counseling program
  Interventions: Behavioral: Tri-focal cognitive behavioral therapy - social skills training (CBTSS) counseling program
- 2 (Active Comparator): Participants will receive the standard care comparison condition
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Tri-focal cognitive behavioral therapy - social skills training (CBTSS) counseling program — This condition is a Theory-Based Counseling Program. The program will involve nine 90-minute face-to-face counseling sessions that use CBT and strategies associated with social cognitive theory. The theory addresses three treatment domains, including mood regulation, reduction/cessation of meth use, and reduction of high risk sexual practices.
  Arms: 1
Behavioral: Standard care — Standard care involves nine weekly, face-to-face individual counseling sessions that provide standard care in relation to sexual risk, methamphetamine use, and depression. The sexual risk component is a modified version of Project RESPECT 1 (CDC, Atlanta) that focuses on educational materials and personal risk appraisal. The meth component is a modified version of the 12-step drug abstinence program developed by the National Institute of Alcohol Abuse and Alcoholism (NIAAA) (Project MATCH). The depression component is an educational approach based primarily on materials provided by the National Alliance on Mental Illness (NAMI) and the National Institute of Mental Health (NIMH).
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of a sexual risk reduction intervention in reducing sexual risk behavior in HIV uninfected, heterosexual people who use methamphetamine.

DETAILED DESCRIPTION:
Methamphetamine is an addictive stimulant drug that strongly activates certain systems in the brain and can cause strong feelings of euphoria. Methamphetamine use has been associated with high risk sexual practices, such as unprotected anal and vaginal sex, multiple sex partners, and sex with partners who inject drugs. These behaviors and others have led to higher rates of STD- and HIV-infections among methamphetamine users. Despite the connection between methamphetamine use and high risk sexual behaviors, few efforts have been made to develop and implement sexual risk reduction programs for this population. Studies of risk reduction programs for "at risk" populations have shown that longer programs are more effective in maintaining improvements in sexual risk behaviors. This study will evaluate the effectiveness of a long-term sexual risk reduction intervention in reducing sexual risk behavior among heterosexual, HIV uninfected people who use methamphetamine.

Participants in this 12-month, open-label study will be randomly assigned to one of the following two conditions: 1) "Tri-focal Cognitive Behavioral Therapy - Social Skills Training (CBTSS) Counseling Program." This condition represents the active experimental condition. Consistent with the theoretical framework, this condition will involve nine 90-minute face-to-face counseling sessions that use cognitive behavioral therapy and strategies associated with social cognitive theory and the theory or reasoned action to address three treatment domains-mood regulation, reduction/cessation of meth use, and reduction of high risk sexual practices. 2) "Standard Care Comparison Condition." Subjects who are assigned to this condition will participate in nine weekly, face-to-face individual counseling sessions that provide standard care in relation to sexual risk, methamphetamine use, and depression. The sexual risk component is a modified version of Project RESPECT (CDC, Atlanta)1 that focuses on educational materials and personal risk appraisal. The meth component is a modified version of the 12-step drug abstinence program developed by the National Institute of Alcohol Abuse and Alcoholism (NIAAA)(Project MATCH). The depression component is an educational approach based primarily on materials provided by the National Alliance on Mental Illness (NAMI) and the National Institute of Mental Health (NIMH). All three programs are widely available and used in community practice.

ELIGIBILITY:
Inclusion Criteria:

* HIV uninfected
* Use of methamphetamine via snorting or smoking at least once a month for the 2 months prior to study entry
* Heterosexual
* History of unprotected sex within 2 months prior to study entry

Exclusion Criteria:

* Current diagnosis of a major psychiatric disorder with psychotic or suicidal symptoms
* History of consistent use of condoms or dental dams for oral, vaginal, or anal sex with all partners within 2 months prior to study entry
* Currently trying to get pregnant or get a partner pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2006-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Frequency of unprotected oral, anal, or vaginal sex | Measured at Months 4, 8, and 12

SECONDARY OUTCOMES:
Depressive symptoms | Measured at Months 4, 8, and 12
Methamphetamine use | Measured at Months 4, 8, and 12
STI incidence (gonorrhea, Chlamydia) | Measured at Month 12
HIV serostatus | Measured at Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L. Patterson, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- HIV Neurobehavioral Research Center, San Diego, California, United States